CLINICAL TRIAL: NCT07066709
Title: Identifying and Managing Pain Generators in Patients With Persistent Post-hip Arthroscopy Pain Using FDG PET/MRI
Brief Title: Painful Post-Operative Hip Study
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Arthroscopy Association of North America (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025-0271; A536110 (Other: UW Madison); SMPH/ORTHO&REHAB/ORTHO (Other: UW Madison); Protocol Version 6/6/2025 (Other: UW Madison)
Record Dates: First submitted 2025-07-03; First posted 2025-07-15 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-08

CONDITIONS: Unilateral Hip Arthroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Revision hip arthroscopy (Experimental): Participants will have undergone a revision hip arthroscopy and will have a FDG PET/MRI
  Interventions: Combination Product: FDG PET/MRI

INTERVENTIONS:
Combination Product: FDG PET/MRI — Participants will undergo an FDG PET/MRI

SUMMARY:
The goal of this clinical trial is to learn if the hips of people who undergo revision hip arthroscopy look different from the hips of people whose hip pain is resolved with the first hip arthroscopy and of people who choose the steroid injection for pain management.

Participants will complete one PET/MRI scan.

DETAILED DESCRIPTION:
Hip arthroscopy utilization has increased significantly and, as such, people are now dealing with an increase in hip arthroscopy failures. In many cases, a failed hip arthroscopy is treated with a revision hip arthroscopy versus conversion to a total hip replacement, but these procedures may not adequately address the etiology of hip pain in the setting of a failed hip arthroscopy. Physicians need better diagnostic tools to appropriately diagnose post- hip arthroscopy hip pain, so that they can offer the appropriate treatment. The advent of FDG PET/MRI offers a highly sensitive imaging method that detects areas of abnormal inflammation. The sensitivity of this method exceeds that of other imaging modalities (e.g., MRI alone) and gives physicians the best possible chance of detecting abnormal inflammatory or hypermetabolic pathology. The ability to better diagnose pain sources around the articular joint with this unique approach has not yet been explored in the post-arthroscopic hip.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-45
* History of unilateral hip arthroscopy
* Does not have evidence of fracture, infection, or malignancy at 6 months post-hip arthroscopy
* Does not have evidence of depression or other major mental health conditions before the index hip arthroscopy
* Does not have persistent pain that requires opioid use, or does not have a history of opioid abuse
* Does not have any comorbidity results in systemic disease limiting function (ASA physical status classification >3)
* Not currently pregnant
* Presents with persistent pain (≥4/10 on NRS) for at least 6 months post-hip arthroscopy
* Undergo a revision hip arthroscopy with no surgical history on the contralateral limb

Exclusion Criteria:

* No unilateral hip arthroscopy
* Evidence of fracture, infection, or malignancy at 6 months post-hip arthroscopy
* Evidence of depression or other major mental health conditions before the index hip arthroscopy
* Has persistent pain that requires opioid use, or has a history of opioid abuse
* Has any comorbidity results in systemic disease limiting function (ASA physical status classification <3)
* Currently pregnant

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Change in number of lesions | Baseline to 12 months
  Images will be taken using FDG PET/MRI to identify the number of lesions in the hip.
Change in size of lesions | Baseline to 12 months
  Images will be taken using FDG PET/MRI to identify the size of the lesions in the hip.
Change in location of lesions | Baseline to 12 months
  Images will be taken using FDG PET/MRI to identify the location of the lesions in the hip.
Change in pain symptoms | Baseline to 12 months
  Participants will self-report pain level of 0-10, with 0 indicating no pain and 10 being the worst pain imaginable.
Change in PROMIs Global Health score | Baseline to 12 months
  Global Health is a participant-reported outcome measure that assesses an individual's overall physical and mental health, including their perceptions of general health. It comprises 10 items, with four items assessing Global Physical Health and four assessing Global Mental Health, all based on five core PROMIS domains: physical function, pain, fatigue, emotional distress, and social health. The scores, ranging from 0 to 20, represent the individual's perception of their health, with lower scores indicating greater impairment.
Change in Hip Outcome Score (HOS) | Baseline to 12 months
  The HOS is interpreted by evaluating scores on two subscales: Activities of Daily Living (ADL) and Sports. Each subscale is scored out of 100, with higher scores indicating better function. A score of 100 means no difficulty, while 0 indicates significant issues.
  Each item within the subscales is scored on a scale of 0 to 4, where 0 means "unable to do" and 4 means "no difficulty." The individual item scores are summed and then converted to a 0-100 scale.
Change in Modified Harris Hip Score (mHHS) | Baseline to 12 months
  The mHHS is interpreted based on a 0-100 scale, with higher scores indicating better hip function. Scores below 70 are considered poor, 70-79 fair, 80-89 good, and 90-100 excellent. The mHHS focuses on patient-reported pain and function.
Change in International Hip Outcome Tool score (iHOT) | Baseline to 12 months
  The iHOT is a questionnaire used to assess participant-reported outcomes related to hip conditions. It evaluates various aspects of hip health, including symptoms, functional limitations, sports and recreational activities, and social/emotional well-being. Higher scores on the iHOT generally indicate better hip function and quality of life. The iHOT-33 has 33 questions, each scored on a 100-point visual analog scale, with 0 representing the worst possible quality of life and 100 representing the best.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Spiker, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin - Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes